CLINICAL TRIAL: NCT07160803
Title: Research on the Status and Strategies of Migrant Elderly for Social Network Software Use From the Activity Theory
Brief Title: Migrant Elderly's Social Network Use Intervention: An Activity Theory-Based Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Responsible Party: Principal Investigator, Huang Riyu, Master of Science in Nursing, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Huzhou University
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Elderly Migrants; Social Networks

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two parallel groups (intervention vs control). The intervention group received a 12-week social network usage program based on Activity Theory, while the control group participated in routine social activities and received the compensatory intervention after the study. Outcomes were assessed at baseline, post-intervention (12 weeks), and 1-month follow-up.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Community Activities+Intervention Program for Social Network Usage Based on Activity Theory (Experimental)
  Interventions: Other: Intervention Program for Social Network Use Based on Activity Theory
- Routine community activities only (Active Comparator)
  Interventions: Other: Routine community activities only

INTERVENTIONS:
Other: Intervention Program for Social Network Use Based on Activity Theory — The intervention program is structured around a three - phase framework for migrant elderly's social network use: ① triggering motivation and building basic capabilities; ② reinforcing motivation and enhancing advanced capabilities; ③ sustaining motivation and maintaining usage habits. The process involves assessing baseline status (via scales like ASNSUS, eHEALS), implementing phased interventions (teaching WeChat skills, facilitating social connections), and evaluating effectiveness (process and outcome evaluations). The 12 - week program is executed by a team including researchers, community workers, and elderly volunteers.
  Arms: Routine Community Activities+Intervention Program for Social Network Usage Based on Activity Theory
Other: Routine community activities only — After receiving regular community services and management, and understanding the overall situation and needs of the intervention targets, researchers and community managers will conduct a weekly health lecture, an offline social activity involving local elderly people (such as fitness, cultural and entertainment activities, etc.), or a lecture on policies and welfare related to migrant elderly people, etc., and regularly distribute relevant paper materials.
  Arms: Routine community activities only

SUMMARY:
This study aims to construct a social network usage intervention program tailored to the characteristics of mobile elderly people, verify its effectiveness, and provide a reference for expanding the field of community care services, bridging the digital divide among mobile elderly people, and promoting their move towards healthy aging.

DETAILED DESCRIPTION:
This study employed a randomized controlled trial (RCT) design, recruiting migrant elderly from a community in Huzhou City as participants. They were randomly assigned to an intervention group and a control group. The control group (n=30) received routine social activities, with compensatory intervention provided after the experiment. The intervention group (n=31) underwent a scientifically valid and operationally feasible practical intervention program, which was developed based on the questionnaire survey method, experimental method, and semi-structured interview method, guided by the Activity Theory, and lasted for 12 weeks.

Before the intervention, after 12 weeks of intervention, and one month after the intervention concluded, standardized scales were used to assess the levels of proactive social network use, basic psychological needs, social isolation, and e-health literacy, respectively. For data analysis, independent-samples t-tests and Spearman correlation analysis were performed based on data distribution patterns and homogeneity of variance, while multiple linear regression was applied for multivariate analysis. Inter-group comparisons post-intervention utilized two independent-samples t-tests and Mann-Whitney U tests, whereas intra-group comparisons employed paired-samples t-tests and Wilcoxon signed-rank tests. The significance level was set at α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* ① Females aged ≥ 55 years or males aged ≥ 60 years; ② Having resided for more than half a year; ③ Having agreed to participate in this study and signed the informed consent form.

Exclusion Criteria:

* ① Elderly individuals with mental illness or cognitive impairment; ② Those with severe language communication barriers.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
Active Social Network Sites Use Scale(ASNSUS) | Baseline, immediately after the end of the intervention (Week 12), 1 month after the end of the intervention (Week 16)
  It consists of 4 items, which are answered in a self-report format and scored on a 5-point Likert scale. The scale assesses the frequency with which individuals update statuses, post photos, leave comments, and initiate messages on social networking sites. It has been validated that the Cronbach's alpha of this scale is 0.71. In the present study, the Cronbach's alpha of this scale was 0.72.

SECONDARY OUTCOMES:
Lubben-6 Scale | Baseline, immediately after the end of the intervention (Week 12), 1 month after the end of the intervention (Week 16)
  This scale was developed by American scholar Lubben [80] in 2006. It includes two dimensions: family and friends, with a total of 6 items, using a 5-point Likert scale. If the total score is lower than 12 points, it indicates the existence of social isolation. The lower the score, the greater the risk of social isolation faced by the individual. This scale is currently the most widely used tool for measuring social isolation in the elderly. Its applicability has been verified by many domestic scholars [81], with a Cronbach's alpha coefficient of 0.84. In this study, the Cronbach's alpha coefficient of this scale is 0.80.
Basic Psychological Needs Scale, BPNS | Baseline, immediately after the end of the intervention (Week 12), 1 month after the end of the intervention (Week 16)
  Sheldon et al. developed this scale in 2006, which was later revised in Chinese and verified to be applicable to the elderly population. The revised scale consists of nine items, divided into three subscales: autonomy needs, competence needs, and relatedness needs. A 5-point Likert scale is used, where a higher score indicates a higher level of need satisfaction. It has been verified that the Cronbach's alpha coefficient is 0.90. The Cronbach's alpha coefficient of this scale is 0.88.
eHealth Literacy Scale, (eHEALS) | Baseline, immediately after the end of the intervention (Week 12), 1 month after the end of the intervention (Week 16)
  The eHEALS scale, designed by scholar Norman and others, aims to quantify an individual's skill level in obtaining and applying online health information. In 2013, Guo Shuaijun and others introduced it into China. The Chinese version is a single-dimensional scale. The eHEALS consists of 8 items, and a higher score indicates a higher level of an individual's eHealth literacy. The scale has been tested by many scholars and proven to be applicable to the elderly population, with a Cronbach's alpha coefficient of 0.98. In this study, the Cronbach's alpha coefficient is 0.85.

CONTACTS AND LOCATIONS:
Overall Officials: Meijuan Cao, Study Director — Huzhou University
Locations (1):
- Huzhou University, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No